CLINICAL TRIAL: NCT06162091
Title: Modeling Trajectories of Functional Outcome in Patients With Severe Acquired Brain Injuries Using a Non-Linear Dynamic Evolution Approach.
Brief Title: Modeling Outcome in Patients With Acquired Brain Injuries
Acronym: MOF-ABI
Status: Recruiting | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Istituto S.Anna Crotone (Unknown); IRCCS Centro Neurolesi Bonino Pulejo (Other); Centro Cardinal Ferrari, Fontanellato, Parma (Unknown); Fondazione Istituto G. Giglio, Cefalù (PA) (Unknown); Habilita Istituto di Neuroriabilitazione, Zingonia (BG) (Unknown); Casa Sollievo della Sofferenza IRCCS (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other); Fondazione Salvatore Maugeri (Other); Istituti Clinici Zucchi (Other); Istituto Clinico Humanitas (Other); Istituto Medicina Fisica E Riabilitazione Gervasutta, Udine (Unknown); Montecatone Rehabilitation Institute S.p.A. (Other); Ospedale Di Riabilitazione Fondazione Santa Lucia, Roma (Unknown); Ospedale San Giovanni Battista, Foligno (PG) (Unknown); Ospedale Ss. Trinità Di Fossano, Cuneo (Unknown); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Antonio Cerasa, PhD, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2023-007
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Brain Injuries
Keywords: acquired brain injury; functional outcome; Modeling trajectories; mathematical models
MeSH Terms: conditions — Brain Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with severe acquired brain injuries: Patients with severe acquired brain injuries admitted at intensive Rehabilitation Units for severe acquired brain injury within 3 months from occurrence
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The study will involve at the time of entry into the rehabilitation setting, the collection of data related to demographic and clinical variables assessing:
  1. The Level of responsiveness (Coma Recovery Scale -revised (CRS-r);
  2. Cognitive functioning (Levels of Cognitive Functioning, LCF);
  3. disability (Disability Rating Scale, DRS);
  4. level of care needed (Early Rehabilition Barthel Index, ERBI)
  The Final outcome measure will be the Glasgow Outcome Scale- Extended (GOSE). It will also collect data on clinical variables and presence of medical devices (e.g. decompressive craniectomy, hydrocephalus, tracheostomy, respiration). For all evaluations, two monthly timepoints will be conducted for a total of 12 timepoints until discharge (0 -6 months). If the patient will be hospitalized for more than 6 months, the assessment will be done monthly up to 12 months.

SUMMARY:
Acquired brain injury (ABI) is the leading cause of death and disability worldwide. The degree of severity varies according to a combination of numerous demographics, etiological, clinical, cognitive, behavioral, psychosocial and environmental factors, which can interfere with the effectiveness of rehabilitation interventions and, therefore, with the final outcome.

The most important goal of the modern clinic is to predict in time the progression of possible recovery after the brain injury event in order to provide more effective treatment, but the high heterogeneity and clinical variability and the unpredictability of the onset of comorbidities makes this a hard target to reach.

In recent years, artificial intelligence algorithms have been applied to more precisely define the role of critical variables that can help clinical practice to predict the final outcome. The classical approach of these algorithms provides only probabilistic values on the final outcome, without considering the typology of clinical interventions and overall complications that may appear throughout the hospitalization period.

The objective of this multicentric study is to define a new statistical approach that can describe the dynamics of individual clinical changes occuring during the inpatient intensive rehabilitation care period. The proposed approach combines a principal component analysis (PCA) for dimension reduction (capturing the maximum amount of information and reducing the dimensionality problem) and a nonlinear mathematical modeling for describing the evolution of the clinical course in terms of the resulting new PCA dimensions. By using this approach, we may determine the individual patient's temporal trajectories while examining particular clinical factors. The secondary objective of this study is to validate a new version of the Early Rehabilitation Barthel Index (ERBI), a well-known clinical scale used to measure functional changes in patients with severe acquired brain injury.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical diagnosis of severe acquired brain injury of different etiology (traumatic, hemorrhagic vascular,ischemic vascular, anoxic, infectious, other etiology
* interval since the acute occurrence that led to the clinical condition of ≤3 months duration
* age of 18 years or older
* informed consent signed by family member/caregiver/supporting caregiver

Exclusion Criteria:

* Positive remote medical history of pre-existing disabling neurological or orthopedic conditions and psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe acquired brain injury, of traumatic and no traumatic etiology, within 3 months of the occurrence
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale - Extended | The test needs approximately 5 minutes to complete.
  The Glasgow Outcome Scale - Extended (GOS-E) is a widely used outcome instrument to assess disability and recovery after brain injury. There are 8 categories in the scale: 1 - Dead, 2 - Vegetative State, 3 - Low Severe Disability, 4- Upper Severe Disability, 5- Low Moderate Disability, 6- Upper Moderate Disability, 7- Low Good Recovery and 8-Upper Good Recovery. The minimum score is 1 (dead) and the maximum score is 8 (upper good recovery).

SECONDARY OUTCOMES:
Early Rehabilition Barthel Index | The test needs approximately 20 minutes to complete.
  The Early Rehabilition Barthel Index (ERBI) is usually used to measure functional changes in patients with severe acquired brain injury.
  ERBI consists of 17 items grouped into two sections, A and B. Section A consists of six "negative" items that can be given the scores - 50 and 0, and one item with scores -25 and 0.
  Section B corresponds to the original Barthel Index, with ten "positive" items, with three scores: 0, 5 and 10.
  The total from section A ranges from - 325 to 0 points, the total from section B from 0 to l00. Therefore, the final total, given by A + B, ranges from -325 (the worst) to +l 00 (the best).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cerasa, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panunzi S, Lucca LF, De Tanti A, Cava F, Romoli A, Formisano R, Scarponi F, Estraneo A, Frattini D, Tonin P, Piergentilli I, Pioggia G, De Gaetano A, Cerasa A. Modeling outcome trajectories in patients with acquired brain injury using a non-linear dynamic evolution approach. Sci Rep. 2023 Apr 18;13(1):6295. doi: 10.1038/s41598-023-33560-x. PMID 37072538